CLINICAL TRIAL: NCT05358509
Title: Reducing Anemia in Pregnancy in India: the RAPIDIRON Trial
Acronym: RAPIDIRON
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: Children's Investment Fund Foundation (Other); Jawaharlal Nehru Medical College (Other); S. Nijalingappa Medical College (Unknown); Raichur Institute of Medical Sciences (Unknown); Sawai Mansingh Medical College (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1811-03347
Record Dates: First submitted 2022-04-15; First posted 2022-05-03 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Iron Deficiency Anemia; Infant, Low Birth Weight; Anemia of Pregnancy
Keywords: Anemia; Iron Deficiency Anemia; Intravenous iron; India; Low birth weight infants; Anemia in pregnancy
MeSH Terms: conditions — Anemia, Iron-Deficiency; Anemia | interventions — ferric carboxymaltose; iron isomaltoside 1000; ferric derisomaltose; ferric sulfate

STUDY DESIGN:
Intervention Model Description: 3-arm, randomized-controlled trial involving two intervention arms (two formulations of intravenous iron) and one active, comparator arm (oral iron, standard of care). Pregnant participants will be randomized with a one-to-one-to-one ration to the three study arms.
Masking Description: Oral iron use will not be masked (as tablets will be provided). However, blinding will occur for the two IV iron intervention arms, as participants, primary health center (PHC) staff, and community health center (CHC) infusion teams will only know that participants have been randomly assigned to receive an IV iron infusion without knowing the specific arm and formulation to be used. A pharmacist associated with each CHC performing infusions for the trial will be designated to prepare the randomly assigned IV iron formulation (according to participant weight and manufacturer instructions) on the day of treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- IV iron intervention arm 1 (Experimental): Intervention arm 1 involves a single dose of an IV iron formulation - ferric carboxymaltose - given during pregnancy.
  Interventions: Drug: Ferric carboxymaltose
- IV iron intervention arm 2 (Experimental): Intervention arm 2 involves a single dose of an IV iron formulation - iron isomaltoside - given during pregnancy.
  Interventions: Drug: Iron isomaltoside
- Active comparator (Active Comparator): Participants randomly assigned to the active comparator arm will receive oral iron tablets to take daily, which is the current standard of care.
  Interventions: Drug: Ferric Sulfate

INTERVENTIONS:
Drug: Ferric carboxymaltose — Pregnant participants randomized to intervention arm 1 will receive a single dose of ferric carboxymaltose having 1000mg of iron if they weigh over 50kg. If a participant is under 50kg, they will receive a lower dose as determined by a formula used by the manufacturer (20mg iron/kg body weight). This will be given ideally immediately after randomization, sometime between 14 weeks and 17 weeks of pregnancy.
  Arms: IV iron intervention arm 1
Drug: Iron isomaltoside — Pregnant participants randomized to intervention arm 1 will receive a single dose of iron isomaltoside having 1000mg of iron if they weigh over 50kg. If a participant is under 50kg, they will receive a lower dose as determined by a formula used by the manufacturer (20mg iron/kg body weight). This will be given ideally immediately after randomization, sometime between 14 weeks and 17 weeks of pregnancy.
  Other Names: Ferric derisomaltose
  Arms: IV iron intervention arm 2
Drug: Ferric Sulfate — Pregnant participants randomized to the oral iron arm will be given 200 ferrous sulphate tablets with 60mg elemental iron each, immediately after randomization, and instructed to take two per day (one in the morning and one at night) throughout the remainder of their pregnancy.
  Other Names: Ferric sulphate
  Arms: Active comparator

SUMMARY:
Anemia is a worldwide problem with iron deficiency being the most common cause. When anemia occurs in pregnancy, it increases the risk of adverse maternal, fetal, and postnatal outcomes. Anemia rates are among the highest in South Asia, with a recent national survey indicating that over half of pregnant women in India are classified as anemic. For nearly 40 years, India's first-level treatment for anemia in pregnancy has been oral iron; however, side effects, poor adherence to tablet ingestion, and low therapeutic impact are among reasons to consider a new paradigm for treatment of pregnant women with iron deficiency anemia (IDA). Reducing Anemia in Pregnancy in India: the RAPIDIRON Trial is a 3-arm, randomized-controlled trial designed to assess if a single dose of an intravenous (IV) iron formulation, administered early in the second trimester of pregnancy for treatment of moderate IDA, will result in a greater proportion of participants in the IV iron arms achieving a normal hemoglobin concentration in the third trimester when compared to participants randomized to receive oral iron. This trial is also designed to test the hypothesis that the low birth weight (LBW) rate for participants randomized to the IV iron arms will be lower when compared to the LBW rate of those randomly assigned to the oral iron arm. The three arms include two IV iron arms (arm 1 - ferric carboxymaltose, arm 2 - iron isomaltoside, also known as ferric derisomaltose) and an active, comparator arm receiving oral iron, which is the standard of care. This study will be conducted in two states in India - Karnataka and Rajasthan. This study supports the overall goals of the Indian Ministry of Health and Family Welfare for pregnancy care; thus, all study participants will be followed according to the Ministry's antenatal care guidelines, and data will be collected through 42 days post-delivery.

(see attached protocol for more detail)

DETAILED DESCRIPTION:
Anemia is a worldwide problem with iron deficiency being the most common cause. When occurring in pregnancy, anemia increases the risk of adverse maternal, fetal and neonatal outcomes, including maternal mortality, preterm and low birth weight (LBW) deliveries, perinatal and neonatal deaths, and long-term developmental sequelae in the surviving offspring. Anemia rates are among the highest in south Asia, and India's latest National Family Health Survey (NFHS-5) for 2019-21 indicates that anemia with hemoglobin (Hb) <11.0 g/dL affects over 50% of pregnant women.

Optimal fetal, neonatal and childhood brain growth and development require adequate iron. However, women with moderate to severe anemia during the late 2nd and early 3rd trimesters of pregnancy are often unable to make up their iron deficit. Thus, despite active transport via the placenta, insufficient iron may be transmitted to the developing fetus with consequent negative sequelae, including long-term neurodevelopmental impairment of the newborn.

For close to 40 years, India's first-level treatment for anemia in pregnancy has been oral iron; however, side effects, poor adherence to tablet ingestion and low therapeutic impact are among reasons for consideration of a new paradigm for treatment of pregnant women with iron deficiency anemia. The Government of India has given high priority to reducing the prevalence of anemia in India, and several initiatives have been directed at this objective. The latest anemia strategy, built on prior strategies and supported by the Ministry of Health and Family Welfare, was presented in a 2018 publication, Anemia Mukt Bharat-Intensified National Iron Plus Initiative. The same overall strategy remains in effect, but a few changes have been made to specific intervention guidelines. The updated guidelines can be viewed online. Notably, this research focuses on pregnant women, one of the population groups targeted by Anemia Mukt Bharat which has the goal of reducing prevalence of anemia among children, adolescents and women in the reproductive age group by 3% a year. The current anemia strategy, supported by the RAPIDIRON Trial, can help facilitate India's efforts to achieve a 2025 Global World Health Assembly target of a 50% reduction of anemia among women of reproductive age.

Reducing Anemia in Pregnancy in India: the RAPIDIRON Trial is a 3-arm, randomized-controlled trial. The study intervention is a single dose of an intravenous (IV) formulation - ferric carboxymaltose in arm 1 or iron isomaltoside (also known as ferric derisomaltose) in arm 2 - administered early in the second trimester of pregnancy for treatment of moderate iron deficiency anemia (IDA). The third arm is an active, comparator arm consisting of oral iron, which is the standard of care. For this trial, approximately 4,320 pregnant women with moderate IDA across four research sites in the Indian states of Karnataka and Rajasthan will be randomized with a one-to-one-to-one ratio to the three study arms.

The two primary hypotheses of this trial are as follows:

1. Pregnant participants with moderate IDA who are randomly assigned to receive IV iron early in their second trimester of pregnancy (in addition to the currently recommended daily dose of folic acid) will have a higher conversion rate to non-anemic status (or Hb ≥ 11g/dL) in the last trimester of pregnancy than pregnant women assigned to an oral iron arm and provided iron and folic acid tablets for anemia treatment; and
2. Pregnant participants assigned to receive IV iron will have a lower rate of low birth weight (LBW) deliveries compared to participants in the oral iron group.

This study will be conducted in primary and community health centers (PHCs, CHCS), hospitals, and birthing facilities located in the four research areas in India - three in Karnataka (Bagalkot, Belagavi, and Raichur), and one in Rajasthan (Jaipur). Participants will be recruited from among pregnant women attending participating PHCs and CHCs for regular antenatal care around 12 weeks of pregnancy. Standard of care for this visit includes blood sample analysis to determine hemoglobin (Hb) level, which will act as a pre-screening tool for this trial. Pregnant women with hemoglobin concentrations <7 g/dL are ineligible for participation and will be referred to a facility for evaluation. Pregnant women with Hb between 7 and 10.4 g/dL will be screened for remaining eligibility criteria, educated about the study, and given the opportunity to consent. If initial eligibility criteria is met and consent is provided, blood will be drawn and transported to a central study hospital to confirm moderate anemia (7 - 9.9 g/dL) and iron deficiency status (serum ferritin <30 ng/mL and/or TSAT <20%). If a potential participant is still eligible based on these laboratory parameters, they will be invited to a subsequent study visit (#2) at one of the associated hospitals for a pregnancy-dating ultrasound to confirm the last of the eligibility criteria. This second visit should occur at about 12-16 weeks of pregnancy. Those eligible after the dating ultrasound will be considered for randomization between 14-17 weeks.

Study visit #3 is intentionally designed to occur between 14-17 weeks of pregnancy to coincide with the antenatal care recommendations of the Ministry of Health and Family Welfare. At this visit, all inclusion and exclusion criteria will be applied to determine final eligibility for continued study participation and randomization. Eligible participants will be randomized at a 1:1:1 ratio to each of the three treatment arms. Randomization will be stratified by enrollment by research area, with the four Indian research areas comprising the four randomization strata. Details of the randomization algorithm and the randomization process will be included in a Randomization Plan developed during the preparatory phase of the study.

All randomized participants will be given a single dose of deworming medication, which government guidelines specify should be taken in the second trimester of pregnancy. Participants assigned to the oral iron arm will receive iron and folic acid tablets consistent with the most recent Anemia Mukt Bharat treatment guidelines for dosage and frequency as found online. Participants assigned to an IV iron arm will receive folic acid tablets in accordance with the recommended daily dosage. IV iron infusions will be scheduled, ideally on the same day as randomization, at a participating CHC (though it can be delayed if necessary as long as it is administered by 17 weeks 0 days of pregnancy).

Both IV iron formulations used in this trial are approved and commercially available in India and have been chosen for use in this study for the following reasons: (1) they allow single-dose infusions of up to 1g of iron; (2) they have proven efficacy and availability in many countries of the world; (3) they are associated with very low rates of adverse events; (4) high quality studies show no difference in severe side effects among available IV iron formulations; and (5) there is greater probability that multiple studies of various single-dose formulations will be instrumental in driving down market prices and lead to public sector pricing and greater utilization. All staff involved in administration of IV iron infusions for this trial will be thoroughly trained to ensure infusions are given consistent with manufacturer labeling instructions, including a recommended observational period subsequent to infusion completion (at least 30 minutes). This time should be sufficient to recognize and appropriately address any drug-related reactions, if they occur, as well as accurately record infusion-related data. Visit #4 only applies to participants who received IV iron treatments - two weeks following an IV iron treatment, they will return to the PHC or CHC to provide a blood sample for analysis for serum phosphate levels.

All participants will return to the PHC or CHC to provide blood samples at visits #5 (20 - 24 weeks of pregnancy), #6 (26-30 weeks of pregnancy) and #7 (30-34 weeks of pregnancy). The timing of these visits are consistent with the Ministry of Health and Family Welfare antenatal visit schedule, and blood sample analysis will allow assessment of changes in hemoglobin levels and iron deficiency status throughout pregnancy.

Visit #8 will occur at delivery/birth. It is expected that many participants will deliver at participating PHCs and CHCs, but some may utilize other birthing facilities in the research areas. For the purpose of this study, participants or someone accompanying them to the birthing facility will be asked to inform a trained mobile team (including a nurse and laboratory technician) that will be expected to report to the facility to ensure completion of data collection essential for this study including: collection of blood from participant prior to delivery; collection of cord blood; measuring weight and length of newborn; recording time between birth and umbilical cord clamping, etc.

The final study visit, #9, will occur about 42 days post-delivery. This will take place at the participant's PHC or CHC and involve blood sample collection as well as administration of a quality of life questionnaire and a survey about breastfeeding practices.

ELIGIBILITY:
Inclusion Criteria for Study Consent for Initial Participation:

* Pregnant women between 18-40 years of age at time of consent that received education about the study and were capable of giving informed consent;
* Hemoglobin concentration of 7 - 10.4 g/dL;
* Expressed intent and expectation of remaining in the designated research area during pregnancy and delivering in a facility in or near the research area and remaining in the area to enable study participant and data collection consistent with the research protocol;
* Expressed willingness that specifically includes agreement to randomization to the standard care study arm (of oral iron) or to one of the two arms involving treatment with single-dose IV iron.

Additional Inclusion Criteria for Randomization and Continued Study Participation:

* Iron deficiency anemia, defined for this study as moderate anemia with hemoglobin concentration level between 7 - 9.9 g/dL, serum transferrin saturation (TSAT) <20%, and/or ferritin <30 ng/mL;
* Presence of a live, singleton, intrauterine fetus and dating ultrasound (at visit #2) that indicates a pregnancy that, at randomization, would be between the beginning of week 14 and prior to 17 weeks 0 days.

Exclusion Criteria:

* Fetal anomaly, if detectable when an initial ultrasound is done to date the pregnancy (subsequent discovery of a fetal anomaly is not viewed as an exclusion criterion);
* History of cardiovascular disease, hemoglobinopathy, or other disease or condition considered a contraindication for treatment, including conditions recommended for exclusion by the manufacturers of oral or IV iron to be used in this study;
* Any condition that, in the opinion of the consenting physician, warrants study exclusion.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4368 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2024-01-21 (Actual)

PRIMARY OUTCOMES:
Return to non-anemic status in the last trimester of pregnancy | 30-34 week antenatal visit or prior to delivery
  Return to non-anemic status, defined as hemoglobin concentration ≥11 g/dL, measured at either a 30-34 week antenatal visit or prior to delivery
Low birth weight (<2500 grams) deliveries | Delivery/birth
  Low birth weight (<2500 grams) deliveries

SECONDARY OUTCOMES:
Changes in hemoglobin concentration by moderate anemia subgroups | 30-34 week antenatal visit or prior to delivery
  Changes in hemoglobin concentration will be analyzed by moderate anemia subgroups according to baseline hemoglobin (i.e., 7-7.9, 8-8.9, and 9-9.9 g/dL)
Changes in transferrin saturation | After randomization to 42 days post-delivery
  Changes in transferrin saturation measured as a ratio of serum iron to total iron-binding capacity (%).
Changes in ferritin | After randomization to 42 days post-delivery
  Changes in ferritin measured in ng/mL.
Changes in offspring hemoglobin measured from cord blood | Delivery/birth
  Changes in offspring hemoglobin concentration from cord blood measured in g/dL
Offspring transferrin saturation from cord blood | Delivery/birth
  Transferrin saturation measured as a ratio of serum iron to total iron-binding capacity (%).
Offspring ferritin from cord blood | Delivery/birth
  Measured in ng/mL.
Weight gain | After randomization to delivery
  Weight gain of participants by trimester of pregnancy
Mode of delivery/incidence of c-section | Delivery/birth
  Mode of delivery, incidence of c-section deliveries
Incidence of hemorrhage | Delivery/birth
  Incidence of antepartum and severe postpartum hemorrhage
Incidence of hypertensive disorders | After randomization to 42 days post-delivery
  Hypertensive disorders
Incidence of maternal infections | After randomization to 42 days post-delivery
  Maternal infections, including documented COVID-19
Incidence of neonatal infections | After randomization to 42 days post-delivery
  Neonatal infections, including documented COVID-19
Incidence of maternal mortality | After randomization to 42 days post-delivery
  Maternal death
Incidence of neonatal mortality | After randomization to 42 days post-delivery
  Neonatal death
Incidence of pregnancy loss and stillbirth | After randomization to delivery
  Pregnancy losses and stillbirths
Newborn length | Measured within 72 hours of delivery
  Birth length of newborns measured in cm
Newborn weight | Measured within 72 hours of delivery
  Birth weight of newborns measured in grams
Incidence of neonatal resuscitation | Within 72 hours of birth
  Neonatal resuscitations
Incidence of neonatal admissions to an intensive care unit | Birth to 28 days of life
  Neonatal admissions to intensive care units within 28 days of delivery
Time from delivery to cord clamping | Within 72 hours of birth
  Time from delivery to umbilical cord clamping
Incidence of unscheduled healthcare visits | After randomization to 42 days post-delivery
  Maternal unscheduled healthcare/hospital visits or extended hospitalizations
Incidence of breastfeeding | 42 days after delivery
  Breastfeeding and exclusive breastfeeding practices, as self-reported by mothers at the 42 day postpartum visit
Well-being/quality of life | 42 days after delivery
  Maternal well-being/quality of life, as measured by the World Health Organization Disability Assessment Schedule II (WHODAS-II)
Incidence of need for 'rescue therapy' | After randomization to delivery
  Incidence of need for 'rescue therapy' or measures implemented for management of severe anemia if a participant's hemoglobin drops below 7 g/dL
Referral for evaluation due to little improvement | 26-30 weeks of pregnancy
  Incidence of referral of a participant, regardless of study arm, to a higher level of care for further investigation of causes of anemia and consideration of possible change in treatment approach due to a <1 g/dL improvement in hemoglobin concentration after at least 2 months from initiation of the randomly assigned treatment, based on analysis of blood drawn at a study monitoring visit at 26-30 weeks of pregnancy
Incidence of preterm and small for gestational age births | Delivery/birth
  Preterm and small for gestational age births

OTHER OUTCOMES:
An independent cost-effectiveness analysis will be conducted by an expert in the field with a background in health economics and the cost-effectiveness of health care interventions. | After randomization to 42 days post-delivery
  This analysis will compare costs of administration of each IV iron formulation used in this study versus oral iron therapy, taking into consideration costs associated with clinical outcomes of IDA in pregnancy.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Derman, MD, MPH, Principal Investigator — Thomas Jefferson University
Locations (4):
- India (4):
  - S. Nijalingappa Medical College, Bagalkot, Karnataka
  - Jawaharlal Nehru Medical College, Belagavi, Karnataka
  - Raichur Institute of Medical Sciences, Rāichūr, Karnataka
  - Sawai Man Singh Medical College, Jaipur, Rajasthan

REFERENCES:
- [Background] International Institute for Population Sciences (IIPS). National Family Health Survey-5, 2019-21, India Fact Sheet. Retrieved 8 February 2022 from: http://rchiips.org/nfhs/NFHS-5_FCTS/India.pdf.
- [Background] Ministry of Health and Family Welfare, Government of India. (April 2018). Anemia Mukt Bharat - Intensified National Iron Plus Initiative (I-NIPI) - Operational Guidelines for Programme Managers. Retrieved 13 April 2022 from: https://anemiamuktbharat.info/wp-content/uploads/2019/09/Anemia-Mukt-Bharat-Operational-Guidelines-FINAL.pdf.
- [Background] electronic medicines compendium (emc). Ferinject (ferric carboxymaltose). Retrieved 30 July 2020 from: https://www.medicines.org.uk/emc/product/5910/.
- [Background] electronic medicines compendium (emc). Monofer 100mg/ml solution for injection/infusion. Retrieved 30 July 2020 from: https://www.medicines.org.uk/emc/product/5676/smpc.
- See also: Anemia Mukt Bharat - India National Anemia Guidelines for Program Managers — https://anemiamuktbharat.info/wp-content/uploads/2019/09/Anemia-Mukt-Bharat-Operational-Guidelines-FINAL.pdf
- See also: Ferinject (ferric carboxymaltose) - Summary of Product Characteristics — https://www.medicines.org.uk/emc/product/5910/
- See also: Monofer 100mg/ml solution for injection/infusion - Summary of Product Characteristics — https://www.medicines.org.uk/emc/product/5676/smpc

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-10): https://cdn.clinicaltrials.gov/large-docs/09/NCT05358509/Prot_SAP_000.pdf